CLINICAL TRIAL: NCT07060534
Title: Building Healthy Eating and Self-Esteem Together for University Students (BEST-U): A Pilot Randomized Controlled Trial of an mHealth Intervention for Binge-Spectrum Disorders
Brief Title: Building Healthy Eating and Self-Esteem Together for University Students
Acronym: BEST-U
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00144380; R34MH134930-01A1 (NIH)
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-06

CONDITIONS: Eating Disorders (Excluding Anorexia Nervosa); Binge-Eating Disorder
Keywords: Eating disorders; Bulimia nervosa; Binge-eating disorder; College Students; Purging disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Bulimia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Present-Centered Therapy (Experimental): PCT is a brief intervention that focuses on building adaptive responses to current life stressors that are directly or indirectly related to psychopathology. PCT focuses on resolving interpersonal disconnection through the development of a positive therapeutic relationship, encouraging connection with others, and addressing interpersonal concerns. We chose PCT as a comparator because it targets daily life stressors, which are important triggers of negative emotions and emotion dysregulation that lead to binge-eating and other eating-disorder symptoms.
  Interventions: Behavioral: Present-Centered Therapy
- BEST-U intervention (Experimental): Building Healthy Eating and Self-Esteem Together for University Students (BEST-U) is a transdiagnostic guided self-help ED treatment for adults that uses evidence-based principles to modify unhelpful thoughts and behaviors that maintain ED and trauma-related psychopathology. The program consists of 15 brief modules delivered each week over 12 sessions. Modules take approximately 10 minutes to complete and focus on key information/lessons that are short and interactive. BEST-U leverages frequent assessment to increase awareness of, and target, problem behaviors. Users reinforce their learning through weekly 25-30-minute telehealth "coaching" sessions, to review module material, problem-solve, practice skills, and plan homework exercises. BEST-U modules and coaching sessions utilize lessons and exercises drawn from Cognitive Behavioral Therapy Enhanced (CBT-E), traditional Cognitive Behavioral Therapy (CBT), and Dialectical Behavior Therapy (DBT).
  Interventions: Behavioral: Building Healthy Eating and Self-Esteem Together for University Students

INTERVENTIONS:
Behavioral: Building Healthy Eating and Self-Esteem Together for University Students — Building Healthy Eating and Self-Esteem Together for University Students (BEST-U) is an mHealth program that includes modules based on second- and third-wave behavior therapy deployed through a smart phone app paired with 20-30-minute coaching sessions. BEST-U incorporates a range of evidence-based skills, and the electronic format allows coaches immediate and easy access to participant reports. BEST-U provides a comprehensive all-in-one assessment and intervention package, is easy-to-implement, brief, and has been tested across genders and in diverse ages and ethnic groups. BEST-U, therefore, has the potential to deliver effective, time-limited, interventions applicable to all university students in routine student healthcare settings.
  Arms: BEST-U intervention
Behavioral: Present-Centered Therapy — Present-Centered Therapy (PCT) is a brief intervention that focuses on building adaptive responses to current life stressors that are directly or indirectly related to psychopathology. PCT focuses on resolving interpersonal disconnection through the development of a positive therapeutic relationship, encouraging connection with others, and addressing interpersonal concerns. PCT was originally developed as a "placebo" intervention for post-traumatic stress disorder but is significantly more efficacious than wait-list in reducing psychiatric symptoms.
  Arms: Present-Centered Therapy

SUMMARY:
Eating disorders (EDs) are a critical concern on college campuses. Moreover, since the COVID-19 pandemic, ED prevalence has increased by 62% in university women and 140% in university men. Resources are inadequate to meet demand, leading to delays in students' access to treatment. Untreated (or poorly treated) EDs result in greater healthcare utilization and costs to students, as well as lower academic achievement and increased psychiatric disability and mortality, suggesting a critical need for quality ED treatment on university campuses and to rethink treatment delivery. One way to address this gap in care delivery is to improve treatment accessibility and scalability, such as dissemination via mobile apps. Guided self-help Cognitive Behavior Therapy (CBT-gsh) is a cost-effective option that can be delivered by non-traditional service providers, such as nurses and physicians. Our scientific premise is that the mHealth CBT-gsh app, Building Healthy Eating and Self-Esteem Together for University Students (BEST-U), will lead to reductions in binge eating (primary outcome) through reductions in dietary restraint and weight/shape concerns (target mechanisms). Prior to implementing BEST-U at other universities, we need to test the intervention in a real-world setting with the end goal of disseminating at scale. Our objectives are to: 1) conduct an effectiveness test of BEST-U compared to a similar dose of present-centered therapy (PCT) in students with non-low weight binge-spectrum EDs and 2) test target mechanisms that lead to changes in binge eating. To accomplish our objectives, we will test the following specific aims: 1) conduct an RCT of BEST-U (N=37) compared to a similar dose of PCT (N=37) in students with non-low weight binge-spectrum EDs; 2) test target mechanisms that lead to changes in binge eating and other ED symptoms; and 3) characterize barriers and facilitators to implementation across two campuses. Our exploratory aim will test food reinforcement and food-choice impulsivity as potential target mechanisms or response moderators of rapid response in binge eating. Given that few studies have identified underlying mechanisms that explain how CBT-gsh works and for whom, this study may lead to improved ability to tailor or modify existing CBT-gsh or lead to novel intervention development for students who are unlikely to respond rapidly (or at all) to first line CBT interventions for EDs.

DETAILED DESCRIPTION:
Eating disorders (EDs) are a critical concern on college campuses and the COVID-19 pandemic has led to increased ED prevalence of 62% in university women and 140% in university men. Resources are inadequate to meet this rising demand as student counseling centers are often understaffed and only 20-21.9% of students reported receiving care for their eating problems, due to financial, logistical, and psychological barriers to accessing treatment. Unfortunately, even when students receive treatment, only a fraction of providers use evidence-based strategies. Untreated (or poorly treated) EDs result in greater healthcare utilization and costs to students, as well as lower academic achievement and increased psychiatric disability and mortality suggesting a critical need for quality ED treatment on university campuses and for rethinking modes of treatment delivery.

One way to address this gap in care delivery is to improve accessibility and scalability of treatment options, such as delivering care via mobile apps. Guided self-help Cognitive-Behavior Therapy (CBT-gsh) is a cost-effective option that can be delivered by a range of non-traditional service providers, such as nurses and physicians. Existing mobile health (mHealth) CBT-gsh programs do not include critical components of CBT such as food and symptom monitoring and reinstatement of regular eating patterns and have limitations that yield low engagement. Our team has developed an easy to use mHealth CBT-gsh program incorporating evidence-based for college students named Building Healthy Eating and Self-Esteem Together for University Students (BEST-U)that includes modules deployed through a smart phone app paired with 20-30 minute coaching sessions. BEST-U incorporates a range of evidence-based skills, and the electronic format allows coaches immediate and easy access to participant reports. BEST-U provides a comprehensive all-in-one assessment and intervention package, is easy-to-implement, brief, and has been tested across genders and in diverse ages and ethnic groups. BEST-U, therefore, has the potential to deliver effective, time-limited, interventions applicable to all young adults in routine student healthcare settings.

Beyond knowing that CBT-gsh interventions are effective generally, it is critical to know how such interventions work and for whom. Without this data, it will remain difficult to: 1) determine what components to add to improve efficacy and 2) identify which clients will respond and which should be referred to alternative care. Thus, novel and scalable treatments to test underlying mechanisms are urgently needed in this population.

Our hypothesis is that the mHealth CBT-gsh app, BEST-U, will lead to reductions in binge eating (primary outcome) through reductions in dietary restraint, weight/shape concerns (targets), and negative emotions. Our pilot data showed strong support for our premise, specifically the need for brief, targeted mHealth interventions in students and the ability of the program to significantly reduce binge eating and impairment and increase wellbeing, with high user acceptability and low drop-out rates. Importantly, these treatment gains were maintained at 3- and 6-month follow-up. However, prior to implementing BEST-U at other universities, we need to test the intervention in a real-world setting with the end goal of disseminating at scale. Thus, we will: 1) conduct an effectiveness test of BEST-U (N=37) compared to a similar dose of present-centered therapy (PCT; N=37) in students with non-low weight binge-spectrum EDs; 2) test target mechanisms that lead to changes in binge eating; and 3) characterize barriers and facilitators to implementing such an intervention across two college campuses.

In addition to our core hypotheses, our exploratory aim is to test food reinforcement and food-choice impulsivity as target mechanisms or response moderators of rapid response in binge eating. Rapid change in binge eating during the first four weeks of CBT-based ED interventions (i.e., "rapid response") is associated with improved end-of-treatment outcomes and aligns temporally with the introduction of "regular eating," a key element for reducing dietary restraint and, thereby, risk for binge eating. However, it is unknown why some individuals respond rapidly to normalization in eating patterns by reducing or eliminating binge eating and why binge eating persists for others. We posit that changes in the relative reinforcement value of food will predict, and food-choice impulsivity will moderate, these differential responses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Student enrolled at KU.
* Bulimia nervosa (BN) or binge-eating disorder (BED) (or sub-threshold BN or BED).
* Access to a smartphone.
* No uncorrected vision problems that would interfere with ability to participate in the study.
* Students taking psychotropic medications must be on a stable therapeutic dose for four weeks prior to study enrollment.
* Able to read and speak fluent English.

Exclusion Criteria:

* Presence of current moderate/severe suicidal ideation with active intent.
* Significant psychopathology that could interfere with treatment (e.g., current substance-use disorder or psychosis).
* Medical conditions or medications that could interfere with treatment (e.g., Type 1 diabetes mellitus, cancer, current pregnancy or nursing, taking corticosteroids, etc.).
* Lab abnormalities indicating medical instability (e.g., low heart rate, electrolyte disturbance, acute medical complications of malnutrition) or another medical problem that would prevent outpatient care as determined through physical health assessment by the student's local clinician.
* Already receiving therapy for an ED.
* Positive screen for anorexia nervosa (AN), atypical AN (AAN), and/or low body weight (i.e., BMI < 19.5) or avoidant and restrictive food intake disorder (ARFID).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-06-23 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Binge eating and total number of eating disorder symptoms measured through the Eating Pathology Symptoms Inventory | Baseline, 12-week intervention (weekly), and 3- and 6-month follow-ups
  The EPSI is a well-validated self-report questionnaire measuring disordered eating symptoms appropriate for use across the weight spectrum and across several demographic groups.
BEST-U Daily Behavior Survey | 12-week intervention (daily)
  Includes self-report of number of daily behaviors, such as binge eating episodes and meal skipping

SECONDARY OUTCOMES:
Clinical Impairment Assessment | Baseline, Week 12, and 3- and 6-month follow-ups
  The Clinical Impairment Assessment is a self-report questionnaire and measures psychosocial impairment secondary to disordered eating concerns.
GAD-7 | Intake, Week 12, 3-month, 6-month follow up.
  The GAD-7 scale is a 7-item questionnaire that assesses how a client has been impacted by symptoms of anxiety over the past two weeks.
PHQ-9 | Intake, Week 12, 3-month follow up, 6-month follow up.
  The Patient Health Questionnaire (PHQ-9) is a nine-item scale used to assess depressive symptoms occurring over the past two weeks in adults.
IDAS-II Dysphoria | Weeks 1-11
  The IDAS-II Dysphoria scale has been shown to correlate strongly with DSM diagnoses of depression (d>1.00), but also has medium to large effect sizes for correlations with panic disorder, posttraumatic stress disorder, and generalized anxiety disorder. Dysphoria also significantly predicts diagnoses of major depression, panic disorder, and generalized anxiety disorder. Assessing Dysphoria on a weekly basis will, therefore, allow us to determine whether changes in negative emotion precede changes in outcomes.

OTHER OUTCOMES:
Body Mass Index (BMI) | Baseline, Weeks 1-12, and 3- and 6-month follow-ups
  Ratio of weight to height
Quick SCID for DSM-5 Disorders | Baseline
  The QuickSCID is a brief, well-validated semi-structured clinical interview of DSM-5-TR disorders. The SCID will be administered to assess lifetime and current DSM-5-TR diagnoses at intake.
EPSI- Clinician Rated Version | Baseline
  The EPSI-Clinician Rated Version (EPSI-CRV) will be administered at intake to obtain a more nuanced assessment of current ED psychopathology.
World Health Organization Disability Assessment Schedule (WHODAS) | Baseline, Week 12; 3-month follow-up; 6-month follow-up
  The WHODAS is a self-report questionnaire measuring general psychiatric impairment and functioning associated with DSM-5 diagnoses.
Inventory of Depression and Anxiety Symptoms (IDAS) | Baseline, Week 12, 3-month follow-up; 6-month follow-up
  Mood and anxiety symptoms and wellbeing will be assessed using the 99-item Inventory of Depression and Anxiety Symptoms (IDAS-II). The IDAS-II has 18 scales and was developed to comprehensively assess internalizing. The IDAS-II has strong internal consistency, inter-rater reliability, and concurrent, discriminant, predictive validity
Computer System Usability Questionnaire (CSUQ) | Week 12
  The Computer System Usability Questionnaire (CSUQ) is a widely used questionnaire that was originally designed to test user satisfaction for computer programs at IBM. The CSUQ has been more recently adapted to assess the acceptability and usability of mHealth apps. Evidence, including our past research, demonstrated that the CSUQ is internally consistent and has a reliable factor structure. In addition to the CSUQ, we will include ad hoc questions that we administered in our pilot study to also inquire about satisfaction with coaching sessions.
Relative reinforcing value of hyper-palatable foods (RRV-HPF) | Weekly (for first 4 weeks)
  Relative reinforcing value of hyper-palatable foods (RRV-HPF) will be measured using a computerized operant behavioral task in which participants will work to earn a preferred (Highly Palatable Food (HPF) or non-HPF alternative. The task assesses food valuation while satiated, to avoid confounding effects of hunger as a motivator. Before beginning the task, participants will choose their most preferred HPF and non-HPF from a list, which will be used in the task. The task requires participants to select which food item they want to earn points for and directs them to work for HPF (or non-HPF). Participants will consume foods as they are earned during the task. After earning a portion of food, the response requirements for another portion of food will be doubled. Participants will be allowed to freely switch back and forth to earn HPF and non-HPF during the task. The task will end when a participant no longer wants to earn the food.
Delay discounting of hyper-palatable foods | Baseline
  A computer-based task will be used to assess choice impulsivity for hyper-palatable foods (HPF), non-HPF, and money. In delay discounting tasks, participants are asked to make a series of choices between a small amount of a reward (e.g., HPF) available immediately, and a larger amount of a reward available at a delay (e.g., HPF in one week). The task will consist of single commodity comparisons between HPF, non-HPF, and money (HPF now vs HPF later; non-HPF now vs non-HPF later; money now vs money later), and cross-commodity conditions that provide choices between one commodity now vs another commodity later (e.g., HPF now vs money later). We will use the following cross-commodity conditions: HPF now vs money later; money now vs HPF later; HPF now vs non-HPF later; non-HPF now vs HPF later.
The Reward-Based Eating Drive Scale-13 (RED-13) | Baseline and 11-week intervention (weekly for first 4 weeks only)
  The Reward-Based Eating Drive Scale-13 (RED-13) measures lack of control overeating, lack of satiety, and preoccupation with food. The RED-13 has excellent psychometric properties and is appropriate to use with the general population and samples with EDs.
The Sensitivity to Reward subscale of the Sensitivity to Punishment and Sensitivity to Reward (SPSRQ) | Baseline and 11-week intervention (weekly for first 4 weeks only)
  The Sensitivity to Reward subscale of the Sensitivity to Punishment and Sensitivity to Reward (SPSRQ) to measure reward sensitivity, and to correlate reward sensitivity with delay discounting for HPF and RRV-HPF.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsie Forbush, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Wakarusa Research Facility, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NIMH requirements, we will share data from the proposed project using the NDA. Data from this project will be preserved to enable sharing through the NDA to validate and replicate the research findings described in our Specific Aims. Data sharing will also enable independent investigators to conduct secondary analyses. Participants will be apprised of how their data will be shared during the consent process. We are committed to sharing research data in a way that is consistent with applicable law and policy, agency mission, and USA national, homeland, and economic security. De-identified data collected from this study will be made publicly available on the NIMH Data Archive. We will restrict any data that may reveal subjects' identities (e.g., geographical location). We view data sharing as crucial for advancing science in eating disorder (ED) research, particularly given that there are few treatment studies of CBT-gsh in young adults.
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: The research community will have access to data when the award ends. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in findability. We will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.